CLINICAL TRIAL: NCT04328571
Title: Effects of Enzymatic Digestion and Probiotic on Oleuropein Bioavailability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 1907NRC
Record Dates: First submitted 2020-03-05; First posted 2020-03-31 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: 3-arms randomized-controlled, parallel group, single center, double-blinded study investigating 3 different formulations of the investigational product
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Single coding
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- OLE enzymatically treated (Experimental): Participants will receive 1 capsule of OLE enzymatically treated + 1 stick of maltodextrin each day in the morning for 21 days
  Interventions: Dietary Supplement: OLE enzymatically treated
- OLE + probiotic (Experimental): Participants will receive 1 capsule of OLE + 1 stick of probiotic each day in the morning for 21 days
  Interventions: Dietary Supplement: OLE + probiotic
- OLE (Active Comparator): Participants will receive 1 capsule of OLE + 1 stick of maltodextrin each day in the morning for 21 days
  Interventions: Dietary Supplement: OLE

INTERVENTIONS:
Dietary Supplement: OLE enzymatically treated — OLE (Olive leaf extract ) enzymatically treated + maltodextrin
  Arms: OLE enzymatically treated
Dietary Supplement: OLE + probiotic — OLE (Olive leaf extract) co-administered with probiotic
  Arms: OLE + probiotic
Dietary Supplement: OLE — OLE (Olive leaf extract) + maltodextrin
  Arms: OLE

SUMMARY:
This is a 3-arms randomized-controlled, parallel group, single center, double-blind study investigating the bioavailability of olive oil extract (OLE) in two different OLE formulations (enzymatically treated and co-administered with a probiotic) compared to original OLE formulation in healthy adult subjects.

DETAILED DESCRIPTION:
Male or female healthy adults between 25 and 65 years of age will be randomized into one of the 3 following groups to receive:

1. Capsule of OLE + 1 stick of maltodextrin
2. Capsule of OLE enzymatically treated + 1 stick of maltodextrin
3. Capsule OLE + 1 stick of probiotic

52 subjects will be randomized to achieve 15 subjects per group to complete the trial.

The study will involve 3 phases:

1. PK1 (all subjects will receive one capsule of OLE in the morning and blood samples will be collected at different timepoints for 24h) followed by a washout period of 1 day
2. 3 weeks intervention (subjects will receive the product thy have benn assigned to) followed by a wash-out period of 3 days
3. PK2 period (subjects will receive one capsule the product thy have benn assigned to

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to sign written informed consent prior to trial entry
2. Male or female healthy adults between 25 and 65 years of age
3. Body Mass Index (BMI) within the range 18.5 - 29.9 (both inclusive)
4. In good health as determined by medical judgment and medical history

Exclusion Criteria:

1. Any food allergy/intolerance
2. Subjects not willing and/or not able to comply with scheduled visits and the requirements of the study protocol
3. Taking or anticipated initiation of any lipid-modifying or blood-clotting medication e.g. statins, cholesterol lowering
4. Smokers
5. Alcohol intake higher than 2 servings per day (one serving is 0.4 dL of strong alcohol, 1 dL of wine, or 3 dL of beer) or drug abuse
6. Receiving or having received antibiotics in the past 4 weeks prior to the day of inclusion
7. Overly imbalanced or restrictive diet (e.g. hyperproteic, vegan, ketogenic, etc.)
8. Hormonal treatment for women linked to menopause (contraceptive treatment accepted)
9. Pregnancy or breastfeeding
10. Supplements or foods containing probiotics (yogurts allowed)
11. Currently participating or having participated in another clinical trial within 4 weeks prior to trial start

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
AUC0-24h of individual blood oleuropein metabolites during PK2 period | 24 hours
  AUC0-24h (concentration/time curve) of individual blood oleuropein metabolites during PK2 period

SECONDARY OUTCOMES:
Cmax during PK2 period | 24 hours
  Cmax of total and individual oleuropein metabolites during PK2 period
Tmax during PK2 period | 24 hours
  Tmax of total and individual oleuropein metabolites during PK2 period
T1/2 during PK2 period | 24 hours
  T1/2 of total and individual oleuropein metabolites during PK2 period
Levels of total and individual oleuropein metabolites in urine at PK2 | 24 hours
  Levels of total and individual oleuropein metabolites excreted in the urine collected over 24 hours during PK2
AUC0-24h during PK1 | 24 hours
  AUC0-24h (concentration/time curve) of individual blood oleuropein metabolites during PK1 period
Cmax during PK1 | 24 hours
  Cmax of total and individual blood oleuropein metabolites during PK1 period
Tmax during PK1 | 24 hours
  Tmax of total and individual blood oleuropein metabolites during PK1 period
T1/2 during PK1 | 24 hours
  T1/2 of total and individual blood oleuropein metabolites during PK1 period
Levels of total and individual oleuropein metabolites in urine at PK1 | 24 hours
  Levels of total and individual oleuropein metabolites excreted in the urine collected over 24 hours during PK1
Change in gut microbiota bacterial population diversity | 3 weeks
  Change from baseline to end of the 3-week intervention period of gut microbiota bacterial population diversity (16SrDNA sequencing)
Change in levels of faecal oleuropein metabolites | 3 weeks
  Change from baseline to end of the 3-week intervention period of faecal oleuropein metabolites

OTHER OUTCOMES:
Change of gut microbiota faecal short chain fatty acids | 3 weeks
  Change from baseline to end of the 3-week intervention period of gut microbiota faecal short chain fatty acids (acetate, propionate, butyrate) & lactate
Change of gut microbiota faecal branched chain fatty acids | 3 weeks
  Change from baseline to end of the 3-week intervention period of gut microbiota faecal branched chain fatty acids (isobutyrate, isovalerate & isocaproate)
Change of gut microbiota faecal ammonium production | 3 weeks
  Change from baseline to end of the 3-week intervention period of gut microbiota faecal ammonium production
Blood levels of total cholesterol | 3 weeks
  Change from baseline to the end of the 3-week intervention period of total cholesterol levels
Blood levels of LDL | 3 weeks
  Change from baseline to the end of the 3-week intervention period of LDL levels
Blood levels of HDL | 3 weeks
  Change from baseline to the end of the 3-week intervention period of HDL levels
Blood levels of ALAT | 3 weeks
  Change from baseline to the end of the 3-week intervention period of ALAT levels
Blood levels of ASAT | 3 weeks
  Change from baseline to the end of the 3-week intervention period of ASAT levels
Blood levels of creatinine | 3 weeks
  Change from baseline to the end of the 3-week intervention period of creatinine levels
Blood levels of glucose | 3 weeks
  Change from baseline to the end of the 3-week intervention period of glucose levels
Blood levels of triglycerides | 3 weeks
  Change from baseline to the end of the 3-week intervention period of triglycerides levels
Blood levels of bone biomarkers | 3 weeks
  Change from baseline to the end of the 3-week intervention period of bone biomarkers (P1NP, CTX)
Blood levels of Oxidized LDL | 3 weeks
  Change from baseline to the end of the 3-week intervention period of Oxidized LDL
Levels of biomarkers of oxidative stress | 3 weeks
  8-NO2GU, 8-OH-GU, 8-OH GUO, 8-OH-DGUO, 8 NO2 GUO, cGMP, 8-NO2-cGMP, Prostanoids, Oxylipins, Isoprostanes, Phytoprostanes and Phytofuranes

CONTACTS AND LOCATIONS:
Overall Officials: Francisco A. Tomás-Barberán, Prof., Principal Investigator — CEBAS-CSIC, Murcia, Spain
Locations (1):
- Universidad Católica San Antonio, Murcia, Spain